CLINICAL TRIAL: NCT00888849
Title: An Open-label, Randomized, Prospective Study of the Effectiveness, Safety, and Clinical Outcomes of Stapled Anastomoses Versus Hand-Sutured Anastomoses in Patients Undergoing Gastrointestinal End to End or Side to Side Anastomoses
Acronym: Tiger
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CI-07-0008
Record Dates: First submitted 2009-04-20; First posted 2009-04-28 (Estimated); Results first posted 2011-11-24 (Estimated); Last update posted 2011-12-05 (Estimated); Status verified 2011-11

CONDITIONS: Gastrointestinal Disease; Colorectal Disease
Keywords: Stapling; hand sutured anastamosis; colorectal disease
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — Sutures

ARMS (2):
- Stapling (Experimental)
  Interventions: Procedure: Advant 55 Linear Cutter/Stapler
- Suturing (Active Comparator): 4 layered hand-sutured anastomosis
  Interventions: Procedure: Suturing

INTERVENTIONS:
Procedure: Advant 55 Linear Cutter/Stapler — Advant 55 Linear Cutter/Stapler
  Arms: Stapling
Procedure: Suturing — Suturing
  Arms: Suturing

SUMMARY:
This study is being conducted to compare surgical and patient outcomes across stapled (Group II) versus hand-sutured (Group I) groups.

ELIGIBILITY:
Inclusion Criteria:a.

* Able to comprehend and sign or, if illiterate, leave their thumb impression on the study informed consent document
* 18 years to 75 years (inclusive)
* Admitted on an emergency or elective basis requiring a single gastrointestinal anastomosis
* Willing to adhere to standard postoperative care, including ventilator support if required
* Female subject is postmenopausal (for at least 2 years) or surgically incapable of child bearing (at least 3 months post-surgical sterilization, with appropriate documentation)
* If female subject is capable of child bearing, must use an acceptable method of birth control (hormonal or IUD) for at least 3 months prior to surgery and continue use throughout the study; maintained normal menstrual pattern for the past three months and has a negative urine pregnancy test prior to day of surgical procedure
* Absence of medical history of psychiatric disorders that could limit the subject's ability to understand the procedure, comply with medical, surgical, and/or behavioral recommendations.

Exclusion Criteria:

* Women of childbearing potential who are pregnant at the time of screening or at the time of surgery
* Subject is on treatment with Corticosteroid maintenance therapy (equivalent to > 10mg/day of Prednisone), immunosuppressive or chemotherapeutic agents within 14 days prior to enrollment; or likely to receive one of these drugs during study period
* Subject has connective tissue disease, renal failure necessitating chronic hemodialysis or chronic ambulatory peritoneal dialysis as evidenced by serum creatinine of > 3mg/dL
* Subject has liver failure as evidenced by CP category C
* Immunocompromised subjects (hematological malignancies, history of bone marrow transplantation, splenectomized subjects, genetic disorders such as Lupus, severe combined immunodeficiency, etc.) or a positive HIV test result
* Subject has extensive disseminated malignancy and unlikely to survive for more than 3 months based on investigator judgment
* Any subject that the investigator determines is not likely to be compliant during the study period
* Subjects determined or suspected to engage in substance abuse, or any subject who is currently, or has in the past 6 months, undergone substance abuse therapy
* The investigator feels that the primary anastomosis is not feasible due to local conditions of the bowel or subject has unstable hemodynamic status requiring stoma
* Participation in any other investigational device or drug study (non survey based trial) within 30 days of enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2009-04; Primary Completion 2010-10 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- India (3):
  - Govt General Hospital and Madras Medical College, Chennai
  - Indira Gandhi Government Medical College, Nagpur
  - GB Pant Hospital, New Delhi

REFERENCES:
- [Background] Choy PY, Bissett IP, Docherty JG, Parry BR, Merrie AE. Stapled versus handsewn methods for ileocolic anastomoses. Cochrane Database Syst Rev. 2007 Jul 18;(3):CD004320. doi: 10.1002/14651858.CD004320.pub2. PMID 17636751

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stapling | Suturing
Started | 142 | 138
Completed | 137 | 129
Not Completed | 5 | 9
Not completed — Death | 4 | 7
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stapling | Suturing | Total
Number analyzed (Participants) | 142 | 138 | 280
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 124 | 128 | 252
  >=65 years | 18 | 10 | 28
Age Continuous [Mean (Standard Deviation); unit: years] | 43.8 (13.81) | 43.7 (15.87) | 43.8 (14.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 56 | 120
  Male | 78 | 82 | 160
Region of Enrollment [Number; unit: participants]
  India | 142 | 138 | 280

OUTCOME MEASURES:

1. Primary Outcome: Time of Surgery (Skin Open to Skin Close)
Time Frame: Day 1
Population: Intent-to-Treat
Measure: Mean (Standard Error); unit: minutes
Groups:
- Suturing: Hand-sutured anastomosis
- Stapling: Stapled Anastomosis
Arm/Group | Suturing | Stapling
Number analyzed (Participants) | 138 | 142
minutes | 168.4 (47.40) | 172.7 (47.40)
Statistical Analysis 1: Comparison: Suturing vs Stapling; Test type: Superiority or Other; p = 0.7774, ANOVA — Adjusted for multiplicity via the Bonferroni-Holm method; Mean Difference (Final Values) = -4.3, 95% CI 2-sided [-19.4 to 10.9], Standard Error of Mean 7.69

2. Primary Outcome: Time of Anastomosis
Time Frame: Total time (minutes) from placement of stay suture to final anastomotic staple (Group II) or final anastomotic suture (Group I)
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Suturing | Stapling
Number analyzed (Participants) | 138 | 142
minutes | 20.6 (1.90) | 17.6 (1.90)
Statistical Analysis 1: Comparison: Suturing vs Stapling; Test type: Superiority or Other; p = 0.0008, ANOVA — Adjusted for multiplicity via Bonferroni-Holm procedure; Mean Difference (Final Values) = 2.9, 95% CI 2-sided [1.4 to 4.5], Standard Error of Mean 0.80

3. Primary Outcome: Return to Bowel Activity
Time Frame: Number of days post-surgery to appearance of peristaltic movement
Measure: Mean (Standard Error); unit: days
Arm/Group | Suturing | Stapling
Number analyzed (Participants) | 138 | 142
days | 4.2 (0.71) | 4.0 (0.71)
Statistical Analysis 1: Comparison: Suturing vs Stapling; Test type: Superiority or Other; p = 0.7774, ANOVA — Adjusted for multiplicity via Bonferroni-Holm procedure; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.2 to 0.6], Standard Error of Mean 0.21

ADVERSE EVENTS:
Arm/Group | Stapling | Suturing
Serious Adverse Events (participants affected / at risk) | 9/142 | 8/138
Other Adverse Events (participants affected / at risk) | 26/142 | 21/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stapling (N=142) | Suturing (N=138)
Bone marrow failure (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Intestinal obstruction (Cardiac disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Wound sepsis (Infections and infestations) | 0 (0) | 1 (1)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Anastomotic fistula (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Failure to anastomose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hemiplegia (Nervous system disorders) | 1 (1) | 0 (0)
Postictal paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stapling (N=142) | Suturing (N=138)
Wound infection (Infections and infestations) | 19 (19) | 11 (11)
Pyrexia (General disorders) | 3 (3) | 6 (6)
Wound secretion (Injury, poisoning and procedural complications) | 6 (6) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other